CLINICAL TRIAL: NCT02204904
Title: A Prospective and Retrospective Data Collection Study to Evaluate Outcomes in Males ≤17 Years of Age Undergoing Allogeneic Hematopoietic Stem Cell Transplantation for the Treatment of Cerebral Adrenoleukodystrophy
Brief Title: Observational Study to Evaluate Allogeneic HSCT Outcomes for Cerebral Adrenoleukodystrophy (CALD)
Status: Terminated | Type: Observational
Why Stopped: Sufficient enrollment for Month 24 safety and efficacy endpoints
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALD-103
Record Dates: First submitted 2014-07-28; First posted 2014-07-31 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2019-12

CONDITIONS: X-Linked Adrenoleukodystrophy (X-ALD); Cerebral Adrenoleukodystrophy (CALD); Adrenoleukodystrophy (ALD)
Keywords: X-linked Adrenoleukodystrophy; Hematopoietic Stem Cells
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Allo-HSCT prospective: Subjects who will be consented before they received an allo-HSC infusion. They will be consented and enrolled on the study during the Screening Period.
  Interventions: Genetic: Allo-HSCT
- Allo-HSCT partial prospective/retrospective: Subjects who will be consented after they received an allo-HSC infusion but before they reach 24 months post-infusion on study. Subjects in this cohort will participate prospectively in at least the Month 24 Visit in order to obtain prospective on-study data for this and all visits after Month 24
  Interventions: Genetic: Allo-HSCT
- Allo-HSCT retrospective: Subjects who received an allo-HSC infusion on or after January 1, 2013 and died before study data collection.
  Interventions: Genetic: Allo-HSCT

INTERVENTIONS:
Genetic: Allo-HSCT — Allogeneic Hematopoietic Stem Cell Transplantation

SUMMARY:
Study ALD-103 will be a multi-site, global, prospective and retrospective data collection study that is designed to evaluate outcomes of allo-HSCT in male subjects with CALD ≤17 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent from a competent custodial parent or guardian with legal capacity to execute a local Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved consent. In addition, informed assent will be sought from capable subjects, in accordance with the directive of the institution's IRB/IEC and all other local requirements.
2. Be male and ≤17 years of age at the time of treatment, for retrospective and partial prospective/retrospective subjects, or at the time of parental/guardian consent and, where appropriate, subject assent, for prospective subjects.
3. Have a confirmed diagnosis of CALD as defined by abnormal VLCFA profile and cerebral lesion on brain MRI.
4. Depending on the cohort, the subject must:

   * Be scheduled for allo-HSCT evaluation at a study site (prospective cohort only),
   * Have received an allo-HSC infusion and be consented in time to complete the Month 24 Visit on study (partial prospective/retrospective cohort only), or
   * Have received their most recent allo-HSC infusion on or after January 1, 2013 (retrospective cohort only).

Exclusion Criteria:

1. Previous treatment with a gene therapy product.
2. Receipt of an experimental transplantation procedure.

Max Age: 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Boys aged 17 or younger receiving allogeneic hematopoietic stem cell transplantation for the treatment of cerebral adrenoleukodystrophy prospectively or partially prospective/retrospective
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Incidence of transplant-related mortality (TRM). | Through 100 and 365 days post allo-HSC infusion
  TRM is defined as death due to any transplantation-related cause other than disease progression.
Incidence and timing of neutrophil engraftment. | 1-48 (± 1) months post allo-HSC infusion
Incidence and timing of platelet engraftment | 1-48 (± 1) months post allo-HSC infusion
Incidence of engraftment failure or allograft rejection. | 1-48 (± 1) months post allo-HSC infusion
Incidence of primary donor-derived chimerism of ≥50%. | by 100 days post allo-HSC infusion
Frequency and severity of Criteria for Adverse Events (CTCAE) ≥Grade 3 AEs, CTCAE ≥Grade 3 infections, and all SAEs. | 1-48 (± 1) months post allo-HSC infusion
Proportion of subjects who experience either ≥Grade II acute (Graft versus Host Disease) GVHD or chronic GVHD. | 1-48 (± 1) months post allo-HSC infusion
Incidence of ≥Grade II acute GVHD. | 1-48 (± 1) months post allo-HSC infusion
Incidence of chronic GVHD. | 1-48 (± 1) months post allo-HSC infusion
Number of emergency room visits. | 1-48 (± 1) months post allo-HSC infusion
Number and duration of intensive care unit stay. | 1-48 (± 1) months post allo-HSC infusion
Number and duration of in-patient hospitalization. | 1-48 (± 1) months post allo-HSC infusion

SECONDARY OUTCOMES:
Incidence of Major Functional Disabilities (MFDs). | 1-48 (± 2) months post allo-HSC infusion
  MFDs is defined as any of the following: loss of communication, cortical blindness, tube feeding, total incontinence, wheelchair dependence, or complete loss of voluntary movement.
Change from Baseline in Loes score | 1-48 (± 2) months post allo-HSC infusion
Change from Baseline in Neurological Function Score (NFS) | 1-48 (± 2) months post allo-HSC infusion
Frequency and timing of resolution of gadolinium enhancement on MRI, if applicable | 1-48 (± 2) months post allo-HSC infusion
MFD-free survival | 48 (± 2) months post allo-HSC infusion
Overall survival | 48 (± 2) months post allo-HSC infusion

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth McNeil, MD MSc, Study Director — bluebird bio, Inc.
Locations (13):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Boston Children's Hospital/Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hospital Austral, Buenos Aires, Argentina
- McGill University Health Centre, Montreal, Quebec, Canada
- University Hospital Leipzig, Leipzig, Germany
- IRCCS Ospedale Pediatrico Bambine Gesú, Roma, Italy
- Princess Maxima Center for Pediatric Oncology (PMC), Utrecht, Netherlands
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chiesa R, Boelens JJ, Duncan CN, Kuhl JS, Sevin C, Kapoor N, Prasad VK, Lindemans CA, Jones SA, Amartino HM, Algeri M, Bunin N, Diaz-de-Heredia C, Loes DJ, Shamir E, Timm A, McNeil E, Dietz AC, Orchard PJ. Variables affecting outcomes after allogeneic hematopoietic stem cell transplant for cerebral adrenoleukodystrophy. Blood Adv. 2022 Mar 8;6(5):1512-1524. doi: 10.1182/bloodadvances.2021005294. PMID 34781360